CLINICAL TRIAL: NCT03352128
Title: The Effect of Creatine Supplementation on Cognitive and Physical Tests
Brief Title: Creatine Supplementation and Cognitive and Physical Tests
Acronym: CREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CREA
Record Dates: First submitted 2017-11-08; First posted 2017-11-24 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Healthy; Creatine Supplementation
MeSH Terms: interventions — Creatine; calcium lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine supplementation (Experimental): 7-day creatine supplementation
  Interventions: Dietary Supplement: Creatine
- Placebo supplementation (Placebo Comparator): 7-day calcium lactate supplementation
  Interventions: Dietary Supplement: Calcium lactate

INTERVENTIONS:
Dietary Supplement: Creatine — Participants will have to supplement themselves with creatine for 7 days (20g/day).
  Arms: Creatine supplementation
Dietary Supplement: Calcium lactate — Participants will have to supplement themselves with calcium lactate for 7 days (elemental calcium: 0.780g/day).
  Arms: Placebo supplementation

SUMMARY:
To assess whether brain creatine availability has an effect on cognition. To do so we will seek to increase brain creatine concentration via a creatine supplementation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological illness including cardiovascular, renal, and endocrine disorder)
* Male/female
* No medication / supplements
* Non-smoker
* Low to moderately active
* Between 18 and 35 years old

Exclusion Criteria:

* Injuries
* Illness
* Use of medication
* Use of creatine in the last 3 months
* History of head trauma or seizure
* Vegetarian diet [24]
* Not being able to follow up the restrictions and prohibitions for the subjects (see Restrictions and prohibitions for the subjects)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Cognitive performance - change in accuracy (%) during a 90-min cognitive task (i.e. Stroop task) | During both lab visits (i.e. after both 7-day supplementation protocols); Accuracy (%) will be assessed during both lab visits with a 90-min cognitive task; Accuracy during the 90-min task will be reported as mean accuracy during 8 blocks of 11min15sec
  Accuracy (in %) will be assessed during a cognitive task, this cognitive task will be completed after both 7-day supplementation protocols (i.e. placebo and creatine)
Cognitive performance - change in reaction time (milliseconds) during a 90-min cognitive task (i.e. Stroop task) | During both lab visits (i.e. after both 7-day supplementation protocols); Reaction time (RT) will be assessed during both lab visits with a 90-min cognitive task; RT during the 90-min task will be reported as mean RT during 8 blocks of 11min15sec
  Reaction time (in milliseconds) will be assessed during a cognitive task, this cognitive task will be completed after both 7-day supplementation protocols (i.e. placebo and creatine)

SECONDARY OUTCOMES:
Physical performance - reaction time (milliseconds) during a 7-min visuomotor reaction time task | During both lab visits (i.e. after both 7-day supplementation protocols); visuomotor reaction time will be assessed during both lab visits with a 7-min visuomotor reaction time task.
  Reaction time (in milliseconds) will be assessed during a visuomotor reaction time task, this physical task will be completed after both 7-day supplementation protocols (i.e. placebo and creatine)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Physiology and Sports Physiotherapy Research Group, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No